CLINICAL TRIAL: NCT07000669
Title: Safety and Efficacy of Bilateral Peribulbar Block for Cataract Surgery
Brief Title: Bilateral Peribulbar Block for Cataract Surgery
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ibrahim Elshahawy, Consultant Anesthesiology, MAGRABI Hospital and Centers, Kingdom of Saudi Arabia, Tanta University
Other Study IDs: 36264PR1192/4/25.
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Safety; Efficacy; Bilateral; Peribulbar Block; Cataract Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peribulbar anesthesia group: Patients undergoing bilateral peribulbar anesthesia for cataract surgery
  Interventions: Other: Bilateral peribulbar block

INTERVENTIONS:
Other: Bilateral peribulbar block — Patients undergoing bilateral peribulbar anesthesia for cataract surgery.

SUMMARY:
This study aims to evaluate the safety and efficacy of bilateral peribulbar block for cataract surgery.

DETAILED DESCRIPTION:
Cataract surgery is one of the most commonly performed procedures worldwide, with local anesthesia being the preferred method due to its safety, efficacy, and cost-effectiveness.

Peribulbar anaesthesia has gained popularity due to its relative efficacy in generating ocular akinesia and anaesthesia with a reduced risk of consequences such as optic nerve damage and globe perforation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Patients undergoing cataract surgery

Exclusion Criteria:

* Infection at the site of the surgery.
* Allergy to any of the used drugs.
* Coagulopathy.
* Posterior staphyloma.
* Bronchial asthma.
* Bradyarrhythmia.
* Pre-existing ocular muscle paresis.
* Neurological deficit.
* Co-existing inflammatory conditions of eye.
* Complicated cataracts.
* Previously operated eyes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This Case series interventional study will be carried out on 50 patients undergoing cataract surgery at Tanta University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | Intraoperatively
  The pain will be evaluated by straightforward questioning using a 3-point scoring method (no pain = 0, discomfort = 1, pain = 2) during the procedure.

SECONDARY OUTCOMES:
Patient satisfaction | 24 hours postoperatively
  The point in time to satisfactory surgical anesthesia will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Grading of Akinesia | Intraoperatively
  Motor block will be assessed by estimation of globe akinesia in the four quadrants, discriminated by the 4 directions of the gaze: lateral, medial, superior, and inferior. A 3- point scoring method will be chosen, in which 0 = akinesia, 1 = incomplete akinesia, and 2 = natural movement, with a total score ranging from 0-8 for the four muscles.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as coughing, vomiting, hypotension, bradycardia, tachycardia, arrhythmias, proptosis, globe puncture, or retrobulbar hemorrhage will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.